CLINICAL TRIAL: NCT00003450
Title: Phase I Trial of Intraperitoneal Adenoviral p53 Gene Therapy in Patients With Advanced Recurrent or Persistent Ovarian Cancer
Brief Title: Gene Therapy in Treating Patients With Advanced Recurrent or Persistent Ovarian Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066481; UTSMC-089733300; NCI-T97-0096
Record Dates: First submitted 1999-11-01; First posted 2003-12-05 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — advexin

INTERVENTIONS:
Biological: Ad5CMV-p53 gene

SUMMARY:
RATIONALE: Inserting the p53 gene into a person's cancer cells may improve the body's ability to fight cancer or make the cancer more sensitive to chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of gene therapy using the p53 gene in treating patients with advanced recurrent or persistent ovarian cancer or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and toxicities of intraperitoneal adenoviral p53 gene therapy in patients with advanced, recurrent, or persistent ovarian carcinoma. II. Evaluate the vector pharmacokinetics and biologic efficacy of gene transfer, gene expression, and cell death in these patients. III. Determine the immunologic response to therapy in these patients.

OUTLINE: This is a dose escalation study of adenoviral p53 gene therapy. Patients undergo removal of ascites, if present, from the peritoneal cavity followed by a bolus infusion of adenovirus p53 once a week for 3 consecutive weeks, followed by a 2 week rest. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients who experience palliative results with at least stable disease may continue treatment weekly without the rest period. Cohorts of 3-6 patients are treated at each level of adenovirus p53. The maximum tolerated dose is defined as the dose level below that at which 2 of 6 patients experience dose limiting toxicity. Patients who receive the MTD without unacceptable toxicity may continue to receive treatment on a weekly basis.

PROJECTED ACCRUAL: Approximately 15-20 patients will be accrued over 16-18 months for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed invasive ovarian epithelial carcinoma or primary peritoneal carcinoma at time of initial laparotomy No histologically confirmed noninvasive ovarian malignancy or low malignant potential tumor or carcinomatosis from other nonovarian or peritoneal sites At least three courses of first-line combination chemotherapy (platinum and paclitaxel) with either persistent or recurrent disease If no treatment with first-line paclitaxel, salvage paclitaxel failure must be documented prior to eligibility Ascites that is cytologically positive for adenocarcinoma or gross evidence of recurrent disease with ascites, or gross recurrent disease with abdominopelvic washing cytologically positive for adenocarcinoma Adequate peritoneal distribution by Technetium 99 scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: GOG 0-2 Life expectancy: Greater than 12 weeks Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT/SGPT no greater than 2.5 times normal No active hepatitis or chronic liver failure Renal: Creatinine no greater than 2 mg/dL Other: Not HIV positive No concurrent immunosuppressive disorders No active systemic infections or active peritonitis Geographically available for follow-up Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior viral based gene therapy treatments or p53 directed vaccines No other prior gene therapy Chemotherapy: See Disease Characteristics At least 4 weeks since chemotherapy No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since radiotherapy No concurrent radiotherapy Surgery: At least 4 weeks since surgery, including surgery for a perforated bowel, bowel anastamosis, colostomy, or ileostomy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Primary Completion 1999-01 (Actual); Study Completion 1999-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Y. Muller, MD, Study Chair — University of New Mexico Cancer Center
Locations (1):
- Simmons Cancer Center - Dallas, Dallas, Texas, United States